CLINICAL TRIAL: NCT01356121
Title: Randomized Controlled Trial Comparing Effects of Sedation for Upper Gastrointestinal Endoscopy With Propofol Versus Midazolam on Psychometric Tests and Critical Flicker Frequency in Cirrhotics
Brief Title: Trial Comparing Sedation for Endoscopy With Propofol Versus Midazolam in Cirrhotics
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Govind Ballabh Pant Hospital (Other Government)
Responsible Party: Prof Barjesh Chander Sharma, G B Pant Hospital New Delhi 110002
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 5289617
Record Dates: First submitted 2011-05-16; First posted 2011-05-19 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-03

CONDITIONS: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Propofol; Midazolam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Midazolam (Active Comparator): Midazolam (0.5-1.0 mg) will be administered in a similar fashion with incremental dosing at intervals of approximately 1-3 min until a level of sedation will be achieved
  Interventions: Drug: Midazolam
- Propofol (Active Comparator): Propofol will be initiated with a 0.5-1 mg/kg i.v. bolus followed by repeated 10-20 mg doses at variable intervals (approximately 15 s, at the discretion of the endoscopist/nurse) until an appropriate level of sedation will be achieved.
  Interventions: Drug: Propofol
- No Sedation (No Intervention): No sedation given in this group

INTERVENTIONS:
Drug: Propofol — Propofol will be initiated with a .5-1 mg/kg i.v. bolus followed by repeated 10-20 mg doses at variable intervals (approximately 15 s, at the discretion of the endoscopist/nurse) until an appropriate level of sedation will be achieved.
  Arms: Propofol
Drug: Midazolam — Midazolam (0.5-1.0 mg) will be administered in a similar fashion with incremental dosing at intervals of approximately 1-3 min until a level of sedation will be achieved
  Other Names: Midazolaam
  Arms: Midazolam

SUMMARY:
To compare effects of sedation for upper gastrointestinal endoscopy with propofol and midazolam on psychometric tests and critical flicker frequency (CFF) in cirrhotics

DETAILED DESCRIPTION:
Upper GI Endoscopy is routinely performed in patients with chronic liver disease to screen for complications related to portal hypertension such as esophageal and gastric varices and portal gastropathy. Sedation is frequently administered to facilitate patient tolerance.Patients with hepatic dysfunction who undergo endoscopy are at increased risk for complications related to sedation.Propofol has a favorable pharmacokinetic profile in comparison with benzodiazepines and opioids, which makes it especially appropriate for sedation in endoscopy.In previous studies cognitive functions were assessed by various paper and pencil tests. However learning affects the paper and pencil tests if repeated at short interval of time.CFF analysis was found to be sensitive and objective in the quantification of low-grade HE, and there is a significant correlation between CFF and the portosystemic encephalopathy syndrome (PHES) battery.Considering this, we designed a prospective randomized controlled study with cirrhotic outpatients to compare effects of sedation for upper gastrointestinal endoscopy with propofol versus midazolam on psychometric tests and critical flicker frequency in cirrhotics

ELIGIBILITY:
Inclusion Criteria:

* Known chronic liver disease (Child-Pugh class A , B or C ) who presented for upper GI endoscopy for routine variceal screening.
* The diagnosis of liver disease will be based on available past history, serological testing, radiological imaging, and liver histology when available.
* Staging of cirrhosis will be determined by MELD score and by Child-Pugh score . All patients will complete a standard preprocedure history and physical examination to establish current degree of encephalopathy and ascites.

Exclusion Criteria:

* Active GI bleeding
* Overt encephalopathy
* Active alcohol intake during the past 6 weeks
* Significant co morbid illness such as heart, respiratory, or renal failure and any neurologic diseases such as alzheimer's disease, parkinson's disease and nonhepatic metabolic encephalopathies.
* Patients with known allergy to sedative
* hepatocellular carcinoma
* Previous TIPS or shunt surgery,
* Patients on psychoactive drugs, such as antidepressants or sedatives
* Patients with an American Society of Anesthesiology (ASA) physical status of class IV or V
* Patients with visual or mental impairment who will unable to complete the psychometric testing or CFF

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-06 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Exacerbation of hepatic encephalopathy | 2 hr

SECONDARY OUTCOMES:
Recovery time | 2 hr
Time to discharge | 2 hr

CONTACTS AND LOCATIONS:
Overall Officials: Barjesh C Sharma, MD,DM, Principal Investigator — Govind Ballabh Pant Hospital
Locations (1):
- Prof Barjesh Chander Sharma, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Agrawal A, Sharma BC, Sharma P, Uppal R, Sarin SK. Randomized controlled trial for endoscopy with propofol versus midazolam on psychometric tests and critical flicker frequency in people with cirrhosis. J Gastroenterol Hepatol. 2012 Nov;27(11):1726-32. doi: 10.1111/j.1440-1746.2012.07231.x. PMID 22861074